CLINICAL TRIAL: NCT01090427
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the of Efficacy and Safety of Ustekinumab in the Treatment of Adolescent Subjects With Moderate to Severe Plaque-type Psoriasis (CADMUS)
Brief Title: A Study of the Safety and Efficacy of Ustekinumab in Adolescent Patients With Psoriasis (CADMUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017053; CNTO1275PSO3006 (Other: Janssen Research & Development, LLC); CADMUS (Other: Janssen Research & Development, LLC); 2009-014368-20 (EudraCT Number); NCT02166203 (obsolete NCT alias)
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Psoriasis
Keywords: Ustekinumab; Injection; CNTO 1275; Stelara; Pediatric psoriasis; Adolescents
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ustekinumab Half-standard Dosage (Experimental): Participants will receive ustekinumab at half the standard dosage at Weeks 0, 4, 16, 28, and 40. In addition, all participants will receive a single SC dose of placebo at Week 12.
  Interventions: Drug: Ustekinumab - Half-Standard Dosage; Other: Placebo
- Ustekinumab Standard Dosage (Experimental): Participants will receive ustekinumab at the standard dosage at Weeks 0, 4, 16, 28, and 40. In addition, all participants will receive a single SC dose of placebo at Week 12.
  Interventions: Drug: Ustekinumab - Standard Dosage; Other: Placebo
- Placebo (Experimental): Participants will receive matching placebo at Week 0 and 4, followed by ustekinumab at half-standard or standard dosage at Weeks 12, 16, 28, and 40.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ustekinumab - Half-Standard Dosage — Ustekinumab 0.375 mg/kg, 22.5 mg, or 45 mg based on body weight, administered subcutaneously (under the skin) at Weeks 0, 4, 16, 28, and 40.
  Arms: Ustekinumab Half-standard Dosage
Drug: Ustekinumab - Standard Dosage — Ustekinumab 0.75 mg/kg, 45 mg, or 90 mg based on body weight administered subcutaneously at Weeks 0, 4, 16, 28, and 40.
  Arms: Ustekinumab Standard Dosage
Other: Placebo — Placebo administered subcutaneously at Weeks 0 and 4 or at Week 12.

SUMMARY:
This is a study of the safety and efficacy of ustekinumab (CNTO 1275) in adolescent patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
This is a randomized (drug assigned by chance), double-blind (a medical research study in which neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled, parallel (a medical research study comparing the response in two or more groups of participants receiving different treatments), multicenter of ustekinumab in adolescent participants with moderate to severe psoriasis. The total duration of study will be 60 weeks. The study will consists of 2 parts; a Screening period and a Treatment period. In treatment period participants will receive either ustekinumab half standard dosage, ustekinumab standard dosage or Placebo. Participants receiving ustekinumab half standard dosage and ustekinumab standard dosage at Week 0, will receive placebo at Week 12 and participants receiving placebo at Week 0 will be randomly assigned to either ustekinumab half standard dosage or ustekinumab standard dosage Weeks 12, 16, 28, and 40. Primarily efficacy will be evaluated by physician's global assessment (PGA) score of cleared or minimal disease. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis with or without psoriatic arthritis (PsA) for at least 6 months
* Are candidates for phototherapy or systemic treatment of psoriasis
* Have screening laboratory test results within the study parameters

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis
* Have used any therapeutic agent targeted at reducing interleukin-12 (IL-12) or interleukin-23 (IL-23), including but not limited to ustekinumab and briakinumab
* Received conventional systemic therapies or phototherapy within the last 4 weeks
* Received biologic therapies within the last 3 months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (50):
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Kitchener, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- France (5):
  - Bordeaux
  - Nantes
  - Nice
  - Saint-Etienne
  - Toulouse
- Germany (7):
  - Berlin
  - Dresden
  - Erlangen
  - Essen
  - Hamburg
  - Kiel
  - Mainz
- Hungary (3):
  - Budapest
  - Debrecen
  - Szeged
- Portugal (4):
  - Braga
  - Lisbon
  - Porto
  - Vila Nova de Gaia
- Russia (6):
  - Korolyov
  - Krasnodar
  - Moscow
  - Rostov-on-Don
  - Saratov
  - Yekaterinburg
- Sweden (2):
  - Linköping
  - Stockholm
- Ukraine (7):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Khmelnitskiy
  - Kiev
  - Simferopol
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (3):
  - Cardiff
  - London
  - York

REFERENCES:
- [Derived] Leu JH, Shiff NJ, Clark M, Bensley K, Lomax KG, Berezny K, Nelson RM, Zhou H, Xu Z. Intravenous Golimumab in Patients with Polyarticular Juvenile Idiopathic Arthritis and Juvenile Psoriatic Arthritis and Subcutaneous Ustekinumab in Patients with Juvenile Psoriatic Arthritis: Extrapolation of Data from Studies in Adults and Adjacent Pediatric Populations. Paediatr Drugs. 2022 Nov;24(6):699-714. doi: 10.1007/s40272-022-00533-y. Epub 2022 Sep 28. PMID 36171515
- [Derived] Landells I, Marano C, Hsu MC, Li S, Zhu Y, Eichenfield LF, Hoeger PH, Menter A, Paller AS, Taieb A, Philipp S, Szapary P, Randazzo B. Ustekinumab in adolescent patients age 12 to 17 years with moderate-to-severe plaque psoriasis: results of the randomized phase 3 CADMUS study. J Am Acad Dermatol. 2015 Oct;73(4):594-603. doi: 10.1016/j.jaad.2015.07.002. Epub 2015 Aug 7. PMID 26259989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 volunteers from 10 countries were randomized and treated in this study.
Pre-assignment Details: A total of 110 participants started and completed the first period in the study (ie, controlled period [CP] and entered the 2nd period (ie, After the Controlled Period [after CP]); however, only 101 of the 110 participants completed the 2nd period (after CP) of the study.
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo Subcutaneous (SC) injections at Week 0 and 4.
- Ustekinumab Half-Standard Dosage (CP): Controlled period (Week 0-12) - Ustekinumab Subcutaneous (SC) injections of 0.375 mg/kg for participants with weight <= 60kg, 22.5 mg for participants with weight > 60 to <= 100kg, and 45 mg for participants with weight > 100kg.
- Ustekinumab Standard Dosage (CP): Controlled period (Week 0-12) - Ustekinumab Subcutaneous (SC) injections of 0.75 mg/kg for participants with weight <= 60kg, 45 mg for participants with weight > 60 to <= 100kg, and 90 mg for participants with weight > 100kg.
- Placebo -> Ustekinumab Half-Standard Dosage (After CP): After Controlled period (Week 12-60) - participants receiving Placebo at Weeks 0 and 4 -> receiving Ustekinumab Half-Standard Dosage at Week 12 and 16 then q12w with the last dose at Week 40.
- Placebo -> Ustekinumab Standard Dosage (After CP): After Controlled period (Week 12-60) - participants receiving Placebo at Weeks 0 and 4 -> receiving Ustekinumab Standard Dosage at Week 12 and 16 then q12wk with last dose at Week 40.
- Ustekinumab Half-Standard Dosage (After CP): After Controlled period (Week 12-60) - participants receiving Ustekinumab Half-Standard Dosage at Weeks 0 and 4 -> receiving Ustekinumab Half-Standard Dosage q12wk with the last dose at Week 40.
- Ustekinumab Standard Dosage (After CP): After Controlled period (Week 12-60) - participants receiving Ustekinumab Standard Dosage at Weeks 0 and 4 -> receiving Ustekinumab Standard Dosage q12wk with last dose at Week 40.
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab Half-Standard Dosage (CP) | Ustekinumab Standard Dosage (CP) | Placebo -> Ustekinumab Half-Standard Dosage (After CP) | Placebo -> Ustekinumab Standard Dosage (After CP) | Ustekinumab Half-Standard Dosage (After CP) | Ustekinumab Standard Dosage (After CP)
Started | 37 | 37 | 36 | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.)
Completed | 37 | 37 | 36 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab Half-Standard Dosage (CP) | Ustekinumab Standard Dosage (CP) | Placebo -> Ustekinumab Half-Standard Dosage (After CP) | Placebo -> Ustekinumab Standard Dosage (After CP) | Ustekinumab Half-Standard Dosage (After CP) | Ustekinumab Standard Dosage (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 19 | 18 | 37 | 36
Completed | 0 | 0 | 0 | 17 | 18 | 32 | 34
Not Completed | 0 | 0 | 0 | 2 | 0 | 5 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received a subcutaneous (SC) injection of Placebo at Weeks 0 and 4 then crossover to ustekinumab half-standard dosage (0.375 mg/kg, 22.5 mg, or 45 mg based on body weight) OR ustekinumab standard dosage (0.75 mg/kg, 45 mg, or 90 mg based on body weight) SC injection at Weeks 12, 16, 28, and 40.
- Ustekinumab Half-Standard Dosage: Participants received ustekinumab subcutaneous (SC) injections (0.375 mg/kg, 22.5 mg, or 45 mg based on body weight) at Weeks 0, 16, 28, and 40. In addition, all participants received a single SC dose of placebo at Week 12.
- Ustekinumab Standard Dosage: Participants received ustekinumab (0.75 mg/kg, 45 mg, or 90 mg based on body weight) subcutaneous (SC) injections at Weeks 0, 4, 16, 28, and 40. In addition, all participants received a single SC dose of placebo at Week 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage | Total
Number analyzed (Participants) | 37 | 37 | 36 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.6 (1.46) | 15.1 (1.7) | 14.8 (1.73) | 15.2 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 20 | 56
  Male | 20 | 18 | 16 | 54
Age [Number; unit: participants]
  12-15 years | 15 | 20 | 20 | 55
  16-17 years | 22 | 17 | 16 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Physician's Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 12
Description: The PGA documents the physician's assessment of the participant's psoriasis status according to the following categories: induration, scaling, and erythema. The participant's psoriasis is assessed as 5-point scale as follows: cleared (0), minimal (1), mild (2), moderate (3), or severe (4); higher score indicates worse disease. The table below shows the percentage of participants who achieved a PGA score of 0 or 1 at Week 12 in each treatment group.
Time Frame: Week 12
Population: The primary efficacy analysis was performed using the all randomized subjects analysis set defined as the population of all participants who were randomized to any treatment group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 37 | 37 | 36
Percentage of Participants | 5.4 | 67.6 | 69.4
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

2. Secondary Outcome: The Percentage of Participants Achieving a Psoriasis Area and Severity Index (PASI) 75 Response at Week 12
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72, with higher scores indicating worse disease. A PASI 75 response is defined as a equal to or greater than (=>) 75% improvement in PASI score from baseline. The table below shows the percentage of participants who achieved a PASI 75 response at Week 12 in each treatment group.
Time Frame: Week 12
Population: The analysis of the PASI 75 response at Week 12 was performed using the all randomized subjects analysis set defined as the population of all participants who were randomized to any treatment group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 37 | 37 | 36
Percentage of Participants | 10.8 | 78.4 | 80.6
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

3. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) Score at Week 12 Compared Between the Placebo Group and the Ustekinumab Treatment Groups
Description: The CDLQI is a dermatology-specific quality of life instrument designed to assess the impact of the disease on a child's quality of life. The CDLQI, a 10-item questionnaire has 4 items response options and a recall period of 1 week. In addition to evaluating overall quality of life, the CDLQI can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, leisure, School or holidays, personal relationships, sleep, and treatment. The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0; the higher the score, the greater impairment in quality of life. The table below shows the mean change in CDLQI score from baseline at Week 12 for each treatment group.
Time Frame: Baseline; Week 12
Population: Evaluable participants for CDLQI are the subsets of all randomized participants with evaluable outcome measurements.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 32 | 35 | 32
Scores on a scale | -1.5 (3.18) | -5.6 (6.43) | -6.7 (5.63)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Test type: Superiority or Other; p = 0.003, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] will be used as factors in the model
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] will be used as factors in the model

4. Secondary Outcome: The Percentage of Participants Achieving a Psoriasis Area and Severity Index (PASI) 90 Response at Week 12 Compared Between the Placebo Group and the Ustekinumab Treatment Groups
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72, with higher scores indicating worse disease. The table below shows the percentage of participants who achieved a PASI 90 response defined as achieving a greater than or equal to (≥) 90% improvement in PASI score from baseline.
Time Frame: Week 12
Population: The analysis of the PASI 90 response at Week 12 was performed using the all randomized subjects analysis set defined as the population of all participants who were randomized to any treatment group.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 37 | 37 | 36
Percentage of Participants | 5.4 | 54.1 | 61.1
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

5. Secondary Outcome: The Percentage of Participants Achieving a Physician's Global Assessment (PGA) Score of Cleared (0) and PGA Score of Mild or Better (<=2) at Week 12
Description: The PGA documents the physician's assessment of the participant's psoriasis status according to the following categories: induration, scaling, and erythema. The participant's psoriasis is assessed as 5-point scale as follows: cleared (0), minimal (1), mild (2), moderate (3), or severe (4); higher score indicates worse disease. The table below shows the percentage of participants who achieved a PGA score of 0 and the percentage of participants who achieved a PGA score of 0, 1, or 2 at Week 12 in each treatment group.
Time Frame: Week 12
Population: Efficacy evaluable subjects defined as the subset of all randomized participants with evaluable outcome measurements.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 37 | 37 | 36
Percentage of participants
  PGA of 0 | 2.7 | 32.4 | 47.2
  PGA of 0, 1, or 2 | 32.4 | 81.1 | 83.3
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PGA of 0; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; PGA of 0; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 3: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PGA of 0, 1, or 2; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 4: Comparison: Placebo vs Ustekinumab Standard Dosage; PGA of 0, 1, or 2; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

6. Secondary Outcome: The Percentage of Participants Who Were PASI 50 Responders and the Percentage of Participants With a PASI Score of 0 at Week 12
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). The table below shows the percentage of participants in each treatment group who were PASI 50 responders at Week 12 defined as participants who achieved a greater than or equal to (>=) 50% improvement in PASI score from baseline as well as the percentage of participants with a PASI score of 0.
Time Frame: Week 12
Population: Efficacy evaluable subjects defined as the subset of all randomized participants with evaluable outcome measurements.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 37 | 37 | 36
Percentage of participants
  PASI 50 responders | 29.7 | 81.1 | 88.9
  Participants with PASI score of 0 | 2.7 | 21.6 | 38.9
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PASI 50 responders; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; PASI 50 responders; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 3: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Participants with PASI score of 0; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 4: Comparison: Placebo vs Ustekinumab Standard Dosage; Participants with PASI score of 0; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

7. Secondary Outcome: The Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Total Scale Score, Psychosocial Health Summary Score, and Physical Health Summary Score at Week 12
Description: The PedsQL is a general health-related quality of life measure developed for use in children and adolescent populations. The Generic Core Scale contains 23 items and is comprised of 4 domains: physical, social, emotional, and school functioning. Each domain can be scored independently. Additionally, a Psychosocial Health and Physical Health Summary Score can be calculated as well as a total score. The measure distinguishes between healthy children and children with acute and chronic health conditions and disease severity within a chronic health condition. The measure is applicable for healthy school and community populations, as well as with pediatric populations with acute and chronic health conditions and has versions for both parent and teen report. Scores range from 0 to 100, and higher scores indicate better health related quality of life.
Time Frame: Week 12
Population: Efficacy evaluable subjects defined as the subset of all randomized participants with evaluable outcome measurements available.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 36 | 36 | 36
Scores on a scale
  PedsQL Total scale score | 3.35 (10.044) | 10.81 (12.882) | 8.03 (10.436)
  PedsQL Psychosocial health summary score | 3.66 (9.610) | 12.13 (15.153) | 8.43 (11.812)
  PedsQL Physical health summary score | 2.86 (12.860) | 8.33 (11.378) | 7.29 (13.446)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PedsQL Total Scale Score; Test type: Superiority or Other; p = 0.003, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; PedsQL Total Scale Score; Test type: Superiority or Other; p = 0.028, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model
Statistical Analysis 3: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PedsQL Psychosocial health summary score; Test type: Superiority or Other; p = 0.005, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model
Statistical Analysis 4: Comparison: Placebo vs Ustekinumab Standard Dosage; PedsQL Psychosocial health summary score; Test type: Superiority or Other; p = 0.063, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model
Statistical Analysis 5: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; PedsQL Physical health summary score; Test type: Superiority or Other; p = 0.007, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model
Statistical Analysis 6: Comparison: Placebo vs Ustekinumab Standard Dosage; PedsQL Physical health summary score; Test type: Superiority or Other; p = 0.020, ANOVA on van der Waerden normal Score; Treatment and baseline weight [less than or equal to 60 kg vs greater than 60 kg] were used as factors in the model

8. Secondary Outcome: The Percentage of Participants With CDLQI Scores of 0 or 1 at Week 12 for Randomized Participants With a Baseline CDLQI Score > 1
Time Frame: Week 12
Population: Efficacy evaluable subjects defined as the subset of all randomized participants with evaluable outcome measurements. In addition, this analysis was limited to participants with a CDLQI of 0 or 1 at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab Half-Standard Dosage | Ustekinumab Standard Dosage
Number analyzed (Participants) | 30 | 31 | 30
Percentage of participants | 13.3 | 38.7 | 56.7
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab Half-Standard Dosage; Test type: Superiority or Other; p = 0.027, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Standard Dosage; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (less than or equal to 60 kg vs greater than 60 kg)

ADVERSE EVENTS:
Time Frame: Through Week 60
Description: Adverse events are provided in the tables below for the 110 participants during 2 time periods in the study: during Weeks 0-12 and during Weeks 12-60.
Arm/Group | Placebo (CP) | Ustekinumab Half-Standard Dosage (CP) | Ustekinumab Standard Dosage (CP) | Placebo -> Ustekinumab Half-Standard Dosage (After CP) | Placebo -> Ustekinumab Standard Dosage (After CP) | Ustekinumab Half-Standard Dosage (After CP) | Ustekinumab Standard Dosage (After CP)
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/37 | 0/36 | 0/19 | 0/18 | 5/37 | 1/36
Other Adverse Events (participants affected / at risk) | 17/37 | 15/37 | 13/36 | 15/19 | 13/18 | 28/37 | 23/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=37) | Ustekinumab Half-Standard Dosage (CP) (N=37) | Ustekinumab Standard Dosage (CP) (N=36) | Placebo -> Ustekinumab Half-Standard Dosage (After CP) (N=19) | Placebo -> Ustekinumab Standard Dosage (After CP) (N=18) | Ustekinumab Half-Standard Dosage (After CP) (N=37) | Ustekinumab Standard Dosage (After CP) (N=36)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=37) | Ustekinumab Half-Standard Dosage (CP) (N=37) | Ustekinumab Standard Dosage (CP) (N=36) | Placebo -> Ustekinumab Half-Standard Dosage (After CP) (N=19) | Placebo -> Ustekinumab Standard Dosage (After CP) (N=18) | Ustekinumab Half-Standard Dosage (After CP) (N=37) | Ustekinumab Standard Dosage (After CP) (N=36)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lip Oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Deposit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Bacterial Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 5 | 1 | 5 | 10 | 11 | 11
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 2 | 2
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxoplasmosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 3 | 2 | 3 | 4 | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haematocrit Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph Node Palpable (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 3 | 2 | 3 | 9 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 3
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 3 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 3 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.